CLINICAL TRIAL: NCT03436719
Title: Randomized Controlled Trial of Antibiotic Prophylaxis in Rectal Cancer Surgery: Oral With Intravenous Versus Intravenous Antibiotics.
Brief Title: Antibiotic Prophylaxis in Rectal Cancer Surgery: Oral With Intravenous Versus Intravenous Antibiotics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Rybakov Evgeny, MD, Dr. Med. Sc. State Scientific Centre of Coloproctology, Head of Surgical department of oncoproctology, Moscow, Russian Federation, State Scientific Centre of Coloproctology, Russian Federation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 76
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Rectal Cancer
Keywords: Surgical Site Infection; Rectal Cancer Surgery; Oral Antibiotic; Antibiotic Prophylaxis
MeSH Terms: conditions — Rectal Neoplasms; Surgical Wound Infection | interventions — Anti-Bacterial Agents; Metronidazole; Erythromycin; Cefoperazone; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral with Intravenous (Experimental): Oral metronidazole and erythromycine administration on the day before surgery with intravenous cefoperazone before surgery (30-90 min) and additional doses every third hour during surgery
  Interventions: Drug: Oral antibiotic; Drug: Intravenous antibiotic; Drug: Mechanical Bowel Preparation
- Intravenous (Active Comparator): Intravenous dose cefoperazone before surgery (30-90 min) and additional doses every third hour during surgery
  Interventions: Drug: Intravenous antibiotic; Drug: Mechanical Bowel Preparation

INTERVENTIONS:
Drug: Oral antibiotic — Metronidazole - 500 mg and Erythromycin - 500 mg per os *3 times at 5 p.m.; 8 p.m., 11 p.m. in a day before surgery
  Other Names: Metronidazole; Erythromycin
  Arms: Oral with Intravenous
Drug: Intravenous antibiotic — Cefoperazone - 1000 mg intravenously for 30-90 minutes before surgery
  Other Names: Cefoperazone
Drug: Mechanical Bowel Preparation — Beginning of MBP at 4 p.m. in a day before surgery
  Other Names: polyethylene glycol

SUMMARY:
This is a randomized, controlled, parallel study to determine the efficiency of oral antibiotics in reduction of surgical site infection (SSI) in rectal cancer surgery.

DETAILED DESCRIPTION:
Patients undergoing rectal cancer surgery in a single centre will assigned randomly to combined preoperative oral antibiotics (metronidazole and erythromycin) and perioperative intravenous antibiotics (cefmetazole) (oral+intravenous group) or to perioperative intravenous antibiotics (cefmetazole) alone (intravenous group). The primary endpoint is the overall rate of SSI.

ELIGIBILITY:
Inclusion Criteria:

* Have a planned of resection of rectum
* Have signed approved informed consent form for the study.

Exclusion Criteria:

* Significant simultaneous surgical procedure (e.g., liver resection of metastasis)
* Bacterial infection at the time of surgery or antimicrobial therapy up to 4 weeks before surgery
* Preoperative severe impairment in renal function (creatinine clearance (MDRD) < 30 ml/min)
* Allergy on the study drugs .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Surgical Site Infection | 0 to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No